CLINICAL TRIAL: NCT05011344
Title: Evolution of Protective Immunization Against SARS-CoV-2 Among Hospital Workers in Health Care Facilities
Brief Title: Evolution of Protective Immunization Against COVID-19 Among Hospital Workers in Health Care Facilities
Acronym: ICONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020-39
Record Dates: First submitted 2021-08-09; First posted 2021-08-18 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: serology; healthcare workers
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposed hospital staff (Experimental): Hospital health care or non-health care staff willing to participate in the study:
  * Healthcare personnel (physician, nurse, caregiver) who have worked for a minimum of 2 weeks since March 1, 2020 in a care unit dedicated to the management of patients confirmed or suspected of COVID-19 infection, in the participating centers: intensive care units, emergency rooms, radiology, COVID-19 units;
  * Staff (physician, technician) who have worked for a minimum of 2 weeks since March 1, 2020 in the AP-HM laboratories handling samples from patients confirmed or suspected of having COVID-19 infection.
  Interventions: Other: Blood sample
- 'Non-exposed' hospital workers (Other): Hospital health care worker (physician, nurse, caregiver) willing to participate in the study who has not worked since March 1, 2020 in an intensive care unit or emergency department or other department dedicated to the management of patients confirmed or suspected of having COVID-19 infection.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Seroneutralization and Elisa tests

SUMMARY:
To measure the immunization rate (seroneutralization) in a population of exposed hospital workers (nursing staff assigned to dedicated COVID-19 care units, laboratory staff handling COVID-19 samples).

DETAILED DESCRIPTION:
Current studies on seroconversion and the time course of immunity following exposure to SARS-CoV-2 do not document: i) Seroconversion in populations in repeated and frequent contact with patients; ii) The temporal dynamics of seroconversion at medium term. These two elements are however fundamental in the comprehension and management of this epidemic or of its potential resurgence in the following months and years.

Objective: To measure the immunization rate (seroneutralization) in a population of exposed hospital workers (nursing staff assigned to dedicated COVID-19 care units, laboratory staff handling COVID-19 samples).

Secondary objectives:

1. Determine the kinetics of the protective response over 12 months (4 times).
2. Compare immunization profiles according to: gender, age, lockdown, blood type, occupational class, exposure, asymptomatic/symptomatic.
3. Compare immunization kinetics between exposed and low-exposure hospital workers.
4. To determine the characteristics of the ELISA test in comparison with the reference test (seroneutralization).

Perspectives

* To provide a reliable, affordable and faster serological test.
* Understanding of the natural evolution of seroprotection in a population over time.
* Sensitization to plasma donation for seropositive patients.

ELIGIBILITY:
Inclusion Criteria:

Cohort of exposed hospital workers

- Hospital caregiver or non-clinician agreeing to participate in the study defined as: Healthcare personnel (physician, nurse, orderly, physical therapist, midwives) who have worked for a minimum of 2 weeks since March 1, 2020 in a care unit dedicated to the management of patients confirmed or suspected of COVID-19 infection, in the participating centers: intensive care units, emergency rooms, COVID-19 units;

* Staff (physician, technician) who have worked for a minimum of 2 weeks since March 1, 2020 in the AP-HM laboratories handling samples from patients confirmed or suspected of having COVID-19 infection
* Person affiliated to a social security system

Cohort of 'unexposed' hospital workers

* Hospital care worker (physician, nurse, orderly) willing to participate in the study who has not worked since March 1, 2020 in an intensive care unit or emergency department or other department dedicated to the management of patients confirmed or suspected of having COVID-19 infection.
* Person affiliated with a social security system

Exclusion Criteria:

* Hospital worker declining to participate If the hospital worker changes assignment after the first collection, he/she remains in the exposed cohort.
* Protected adult
* Person under legal guardianship or curatorship

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
To establish the level of immunization (seroprevalence) to COVID-19 as determined by the seroneutralization test in a population of exposed hospital workers | 4, 8 and 12 months follow-up visits after the initial visit
  Positive seroneutralization test result: the threshold of positivity is set at 40, i.e. any serum with a seroneutralizing value greater than or equal to 40 will be considered positive.

SECONDARY OUTCOMES:
Kinetics of the protective antibody immune response (protective immunization against SARS-CoV-2 COVID-19) in a population of exposed hospital workers over a 12-month period. | 4, 8 and 12 months follow-up visits after the initial visit
  The kinetics of "seroprevalence" will be defined by the results of the seroneutralization test at 4 time-points (4, 8 and 12 month follow-up visits after the initial visit).
Compare immunization profiles | 12 months after the initial visit
  Combine multiple measurement in order to compare immunization profiles (symptomatic status,individual characteristics, i.e, gender, age range, condition of lockdown, blood type; professional characteristics and possible clinical signs.
Compare the seroprevalence of SARS-CoV-2 and the kinetics of immunization between two groups (exposed hospital workers and a less exposed hospital workers). | 4, 8 and 12 months follow-up visits after the initial visit
  Compare between groups the results of the seroneutralization test over time.
Identify the technical (sensitivity and specificity) and predictive (positive and negative predictive values) characteristics of the ELISA test evaluated in comparison with the reference test (serum neutralization) in the population of interest. | 12 months
  ELISA's test positivity will be defined with reference to the manufacturer's recommendations. For a ratio OD of the tested sample / kit control:
  * <0.9: negative test
  * Between 0.9 and 1.1: unspecified test
  * >1.1: positive test The result will be processed under two modalities: negative/indeterminate/positive and quantitative
Record COVID-19 seroprevalences established by ELISA at different time points: inclusion, 4 months, 8 months, and 12 months after inclusion. | 4, 8 and 12 months follow-up visits after the initial visit
  The technical and predictive characteristics of the ELISA test (sensitivity, specificity, positive predictive value and negative predictive value) are documented by reference to the serum neutralisation test.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO-PRADALIE, MD, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, France